CLINICAL TRIAL: NCT04780126
Title: Measuring the Loss of Skeletal Muscle Mass in the Hospitalized Patient With the Diagnosis of COVID-19
Brief Title: Sarco-COVID Study: Measuring the Loss of Skeletal Muscle Mass in the Hospitalized Patient With the Diagnosis of COVID-19
Acronym: SARCO-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Principal Investigator, Yale Tung Chen, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Other Study IDs: 21/090-E_COVID
Record Dates: First submitted 2021-02-19; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia; Covid19
Keywords: sarcopenia; covid19
MeSH Terms: conditions — Sarcopenia; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 pneumonia patients: Patients over 18 years of age who are admitted to the hospital and whose main diagnosis and reason for staying is COVID-19 pneumonia will be included.
  Interventions: Other: Sarcopenia diagnosis

INTERVENTIONS:
Other: Sarcopenia diagnosis — History, physical, laboratory and ultrasound parameters to diagnose sarcopenia

SUMMARY:
The COVID-19 pandemic is having a devastating global impact, and older adults who experience it are at higher risk of death from the disease. However, survivors of the disease have a greater risk of suffering from pathologies such as sarcopenia, which is more frequent in younger adults and with greater severity of the disease.

Sarcopenia is present in 5-13% of people between 60 and 70 years old and in 11-50% of the population over 80 years of age. The diagnosis of sarcopenia has advanced in recent years by establishing homogeneous criteria in different consensuses that necessarily combine two elements: generalized loss of strength accompanied by loss of skeletal muscle mass. Today there are three consensuses for the diagnosis of sarcopenia: the international (IWGS), the European (EWGSOP), and the most recent from a US cohort (FNIH). In all of them, the measurement of skeletal muscle mass constitutes one of the two diagnostic criteria.

The main methods to measure this muscle loss that are established are imaging techniques (computerized tomography (CT), magnetic resonance imaging (MRI), dual-energy X-ray absorptiometry (DEXA) and ultrasound.

The most common ultrasound measurements used for this purpose are the muscle thickness (cm) at the point of the ultrasound path of maximum muscle thickness, the cross-sectional area (area calculated by the basic software at the point of maximum muscle thickness), and the pennation angle (angle formed between deep muscle fascia and muscle fibers). The first two measurements can be made on several long muscles, while the pennation angle is usually made primarily on the medial gastrocnemius (internal twin) muscle. They are easy to obtain, bloodless, and reproducible measurements.

Research efforts at this point in the pandemic should focus on the longer-term consequences of the disease, sequelae such as sarcopenia in patients who have suffered from COVID-19. At the same time, clinicians must become increasingly aware of the condition and its measurement integrated into clinical practice. The knowledge provided by studies such as the one presented will allow the development of specific interventions.

The risk of sarcopenia should be considered when carrying out a risk / benefit assessment of the established treatment (for example, dexamethasone), and considering a multidisciplinary treatment that includes dietary inputs.

DETAILED DESCRIPTION:
Patients over 18 years of age who are admitted to the hospital and whose main diagnosis and reason for staying is COVID-19 pneumonia will be included. The prevalence of sarcopenia in hospitalized patients is 15-20%. Assuming an alpha risk of 0.05 and a beta risk of 0.2 in a unilateral contrast, 64 subjects are required to detect a difference equal to or greater than 20% loss of muscle mass. A loss to follow-up rate of 0% has been estimated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, men or women.
* Main diagnosis is pneumonia due to COVID-19
* Subjects who, after having received information about the design, the purposes of the project, the possible risks that may arise from it and who at any time may deny their collaboration, verbally grant their consent to participate in the study.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Present a malignant neoplasm in active phase except spino- or basal cell Ca in local stage
* Clinical situation of agony.
* Amputation of limb (s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who are admitted to the hospital and whose main diagnosis and reason for staying is COVID-19 pneumonia will be included.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Loss of muscle mass | 1 month
  Quantify the loss of muscle mass in hospitalized patients in areas of Internal Medicine with a diagnosis of COVID-19

SECONDARY OUTCOMES:
Prevalence of sarcopenia | 1 month
  Analyze the clinical characteristics and the prevalence of sarcopenia in the patients included in the study.
Normal values of muscle ultrasound thickness | 1 month
  Analyze the thickness of the rectus femoris, vastus medialis, vastus lateralis, medial gastrocnemius in all patients.
C reactive protein (CRP) correlated to the presence of sarcopenia | 1 month
  Analyze the correlation between CRP and the presence of sarcopenia
Therapy with corticosteroids impact on muscle thickness | 1 month
  Determine the correlation between muscle thickness and the corticotherapy received (dexamethasone, methylprednisolone, prednisone)
Normal values of medial gastrocnemius pennation angle in all patients | 1 month
  Measure medial gastrocnemius pennation angle in all patients
Ferritin correlated to the presence of sarcopenia | 1 month
  Analyze the correlation between Ferritin and the presence of sarcopenia
Fibrinogen correlated to the presence of sarcopenia | 1 month
  Analyze the correlation between Fibrinogen and the presence of sarcopenia

CONTACTS AND LOCATIONS:
Overall Officials: Yale Tung Chen, MD PhD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (1):
- Hospital de Emergencias Isabel Zendal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Epidemiologic and methodologic problems in determining nutritional status of older persons. Proceedings of a conference. Albuquerque, New Mexico, October 19-21, 1988. Am J Clin Nutr. 1989 Nov;50(5 Suppl):1121-235. No abstract available. PMID 2816807
- [Result] von Haehling S, Morley JE, Anker SD. An overview of sarcopenia: facts and numbers on prevalence and clinical impact. J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):129-133. doi: 10.1007/s13539-010-0014-2. Epub 2010 Dec 17. PMID 21475695
- [Result] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Result] Fielding RA, Vellas B, Evans WJ, Bhasin S, Morley JE, Newman AB, Abellan van Kan G, Andrieu S, Bauer J, Breuille D, Cederholm T, Chandler J, De Meynard C, Donini L, Harris T, Kannt A, Keime Guibert F, Onder G, Papanicolaou D, Rolland Y, Rooks D, Sieber C, Souhami E, Verlaan S, Zamboni M. Sarcopenia: an undiagnosed condition in older adults. Current consensus definition: prevalence, etiology, and consequences. International working group on sarcopenia. J Am Med Dir Assoc. 2011 May;12(4):249-56. doi: 10.1016/j.jamda.2011.01.003. Epub 2011 Mar 4. PMID 21527165
- [Result] Studenski SA, Peters KW, Alley DE, Cawthon PM, McLean RR, Harris TB, Ferrucci L, Guralnik JM, Fragala MS, Kenny AM, Kiel DP, Kritchevsky SB, Shardell MD, Dam TT, Vassileva MT. The FNIH sarcopenia project: rationale, study description, conference recommendations, and final estimates. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):547-58. doi: 10.1093/gerona/glu010. PMID 24737557
- [Result] Nijholt W, Scafoglieri A, Jager-Wittenaar H, Hobbelen JSM, van der Schans CP. The reliability and validity of ultrasound to quantify muscles in older adults: a systematic review. J Cachexia Sarcopenia Muscle. 2017 Oct;8(5):702-712. doi: 10.1002/jcsm.12210. Epub 2017 Jul 12. PMID 28703496

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT04780126/Prot_SAP_ICF_000.pdf